CLINICAL TRIAL: NCT06705413
Title: Effect of Lifestyle Modification on Obese Females With Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Taha Abd EL-Hamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005311
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Active Comparator): The participants will receive a program of aerobic exercise for 3 consecutive menstrual cycles.
  Interventions: Other: Aerobic exercise
- Aerobic exercise and microbiome diet group (Experimental): The participants will receive aerobic exercise in addition to microbiome diet for 3 consecutive menstrual cycles.
  Interventions: Other: Aerobic exercise; Other: Microbiome diet

INTERVENTIONS:
Other: Aerobic exercise — a program consists of 10 minutes warming up, 30 minutes of aerobic exercises in the form of core strengthening exercises and stretching exercises and finally 10 minutes of cooling down. The participant will receive the aerobic program 4 sessions /week for three consecutive menstrual cycles.
Other: Microbiome diet — The participants will receive Microbiome diet for three consecutive menstrual cycles. A three-phase diet (21-day phase, 28-day phase and maintenance phase) will be followed by the experimental group which contains some food restrictions and addition for certain food types which may improve gut health.
  Arms: Aerobic exercise and microbiome diet group

SUMMARY:
The study will be designed to determine the effect of lifestyle modification on primary dysmenorrhea in obese females.

DETAILED DESCRIPTION:
Menstruation in women after puberty is often confused with dysmenorrhea. Primary dysmenorrhea, where there is no apparent pelvic pathology, is characterized as painful menstrual cramps. This symptom typically occurs within one to two years of menarche and menstrual cycle stabilisation1. Pain occurs a couple of hours before or after menstruation and lasts for 12 to 72 hours. Dysmenorrhea can also be accompanied by nausea, discomfort, low back pain, or flank pain.

Obesity in women adolescents is one of the factors associated with dysmenorrhea also; Endometrium production of physiological prostaglandin increased in primary dysmenorrhea. Increased prostaglandin directly contributes to uterine contractions that eventually lead to primary dysmenorrhea. Overweight and obesity thought to be correlated with dysmenorrhea by increasing the development of prostaglandin.

The Microbiome Diet is a new, trendy weight loss diet. It created by Dr. Raphael Kellman and based on eating and avoiding certain foods in the hopes of restoring gut health. It's also claimed to offer other benefits, such as a faster metabolism and weight loss. Therefore, this study aims to investigate the effect of lifestyle modification on obese females suffering from primary dysmenorrhea

ELIGIBILITY:
Inclusion Criteria:

* Young females with moderate to severe primary dysmenorrhea (Visual analogue scale > 4).
* Virgin, nonsmokers.
* Young female aged from 18-25 years with BMI more than 30 kg/m².
* They have regular menstrual cycles (a menstrual flow of 38 days, with 21-35 days between menstrual flows)
* They have not practiced sports for at least one year before entering the study.
* They have not engaged in diet for at least one year before entering the study.

Exclusion Criteria:

* Any participant having Secondary dysmenorrhea (associated with identifiable pelvic pathology).
* Any participant with a history of pelvic inflammatory disease, myoma and tumors, pelvic infection, ovarian cyst, any gynecological disease.
* Any participant with a history of previous spinal surgeries.
* Any participant with a history of Anemia, diabetes, hypertension, cardiovascular disease, thyroid disease, neurological disorder, rheumatoid arthritis, bariatric surgery, or taking weight loss medication.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 71 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain level assessment | 3 months
  The visual analogue scale will be used to measure menstrual pain intensity for both groups before and after treatment.it is a valid and reliable 10 cm line ranging from 0 to 10. 0 indicates no pain,10 indicates worst pain.
Assessment of severity of dysmenorrhea | 3 months
  WaLIDD scale will be used to determine the severity of dysmenorrhea for each female in both groups by combining subjective (intensity/wong-baker, work ability) and objective (days of pain, location) manifestations for both groups. its score ranges between 0 and 3, and the final score ranges from 0 to 12 points. the higher the score, the greater the severity of dysmenorrhea.
Assessment of pain pressure threshold | 3 months
  the pressure algometer will be used to assess pain pressure threshold for all females in both groups before and after treatment on the following points: A-Two measurements 4cm from the umbilicus, bilaterally (points I and II) B-Two other measurements 4cm below the previous ones (points III and IV) C. A single measurement 4cm from the lower margin of the umbilicus (point V). D. Another single measurement into the medial side of the lumbar region below the fifth lumbar vertebra, corresponding to S2-S4 (point VI).
Body mass index | 3 months
  Weight and height measurement will be measured for each participant in both groups before and after the treatment to calculate her BMI according to the following equation:
  BMI (kg/m2) = Weight (kg) / Height² (m2).
Waist and hip ratio measurement: | 3 months
  Waist hip circumference were taken for each woman in both groups before and after the treatment course for calculating waist and hip ratio (WHR) by dividing the waist circumference (WC) on hip circumference (HC). By the tape measurement, (WC) was measured at the narrowest circumference between xipho-sternum and the iliac crest at the end of gentle expiration. HC was measured at the maximum circumference at the level of femoral trochanter.

SECONDARY OUTCOMES:
Measurement of lumbar mobility | 3 months
  By using the modified Schober test, the participant will be asked to stand; the therapist will mark both posterior superior iliac spines (PSIS) and then will draw a horizontal line connecting the center of both marks. A second line will be marked 5 cm below the first line and a third line will be marked 10 cm above the first line. The participant will be instructed to flex forward as if attempting to touch her toes, then therapist will re-measure the distance between the top and bottom line. The increased distance along the tap due to lumbar flexion is normally about 6-7 cm (less than 5 cm should be considered abnormal)
Measurement of lumbar lordotic curve | 3 months
  The subjects will be asked to stand with lower back and upper buttocks exposed on the markings done by adhesive tape on the floor with a distance of 15 cm between feet.
  The flexible ruler will be placed over the lumbar spinous process and the readings on the flexible ruler that intersected with the markings done on spinous processes will be noted.
  The vertical line (L) will be drawn to connect the spinous processes T12 and S2 landmarks and will be labelled as A and B respectively. The deepest point of the curve will be identified by recording the steep of the curve and a perpendicular line (H) from the point to the line L will be drawn. The L and H lengths will be measured in cm The measurements will be recorded after removing the flexible ruler without changing the curve. Then, the outline of the curve will be traced from the readings for T12 to S2 spinous processes using a pencil along the flexible ruler onto the graph sheet its normal value is ranged between 20° and 45°.
Assessment of Health-Related Quality of Life | 3 months
  It will be assessed before and after treatment program using Free online SF-36 score calculator. The SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). Responses will be scored on a five point scale (from "very poor" to "very good"), where higher scores indicate better enjoyment and satisfaction with life. Scores will be added and presented as a percentage of the total maximum score. A percentage of total score of > 70 represents normal quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa Osman, professor, Study Director — Cairo University; Amel Yousef, Professor, Study Chair — Cairo University
Locations (1):
- Noha Taha Abd El-Hamed, Ismailia, Egypt